CLINICAL TRIAL: NCT03559452
Title: In Young Healthy Males and Females, What is the Effect of Prior Eccentric Exercise on Thigh Muscle Atrophy During One Week of Leg Disuse Compared to no Prior Exercise?
Brief Title: Muscle Damage and Disuse Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 171206/B/08
Record Dates: First submitted 2018-05-31; First posted 2018-06-18 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Muscle Disuse Atrophy
Keywords: Muscle damage; Inflammation; Immobilisation
MeSH Terms: conditions — Muscular Disorders, Atrophic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Immobilisation without prior exercise
- Muscle damage (Experimental): 300 bilateral knee extensor eccentric contraction performed immediately prior to immobilisation
  Interventions: Procedure: Eccentric exercise

INTERVENTIONS:
Procedure: Eccentric exercise — 300 eccentric contractions of the knee extensors
  Arms: Muscle damage

SUMMARY:
Limb injury generally requires a period of recovery during which time the limb is often immobilised (e.g. with a cast or brace) resulting in a rapid loss of skeletal muscle. Despite the importance of muscle loss during injury, our understanding of how it occurs is incomplete. Several factors are likely to contribute, including a lack of muscle contraction and injury induced inflammation. In this study, the investigators will recruit healthy volunteers who will spend 7 days in a knee brace to replicate leg immobilisation. Prior to immobilisation, half of the participants will perform a single session of strenuous resistance exercise which is known to cause muscle damage and initiate an inflammatory response. This is designed to replicate the muscle damage and inflammation that occurs with injury. The remaining half of participants will not perform this exercise, allowing us to look at the additive effect of muscle damage and inflammation on muscle loss with immobilisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 40
* BMI between 18 and 27
* Healthy, recreationally active, non smoker

Exclusion Criteria:

* Non-removable metallic implants (including heart pacemaker, cochlear implants, medication pumps, surgical clips, plates or screws) or claustrophobia
* Use of nutritional supplements
* Chronic use of over the counter medication
* Any diagnosed metabolic disease (e.g. type 1 or 2 Diabetes).
* Any diagnosed cardiovascular disease or hypertension.
* Anyone with previous motor disorders. Anyone with a current musculoskeletal injury that may impair their use of crutches.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in thigh muscle volume from pre-immobilisation | After 2 days of immobilisation
  The volume of the muscles comprising the thigh after 2 days of immobilisation will be compared to pre-immobilisation values. This will be measured using MRI.
Change in thigh muscle volume from pre-immobilisation | After 7 days of immobilisation
  The volume of the muscles comprising the thigh after 7 days of immobilisation will be compared to pre-immobilisation values, and values obtained after 2 days of immobilisation. This will be measured using MRI.

SECONDARY OUTCOMES:
Change in unilateral knee extensor 1 repetition maximum | After 7 days of immobilisation
  Unilateral knee extensor 1 repetition maximum will be measured before and after 7 days of single leg immobilisation using a weight stack leg extension machine
Change in unilateral knee extensor maximal voluntary torque production | After 7 days of immobilisation
  Unilateral knee extensor maximal voluntary torque production will be measured before and after 7 days of single leg immobilisation using an isokinetic dynamometer.
Change in unilateral knee extensor isokinetic total work | After 7 days of immobilisation
  Unilateral knee extensor total isokinetic work after 30 consecutive contractions will be measured before and after 7 days of single leg immobilisation using an isokinetic dynamometer.
Muscle protein synthesis assessed using the stable isotope Deuterium Oxide | After 2 days of immobilisation
  The enrichment of deuterated alanine (from the deuterium oxide heavy water stable isotope tracer) in vastus lateralis biopsy samples will be measured relative to the non-deuterated alanine. The change between pre-immobilisation and 2 days of immobilisation will be used to calculated a fractional synthetic rate (% day).
Muscle protein synthesis assessed using the stable isotope Deuterium Oxide | After 7 days of immobilisation
  The enrichment of deuterated alanine (from the deuterium oxide heavy water stable isotope tracer) in vastus lateralis biopsy samples will be measured relative to the non-deuterated alanine. The change between pre-immobilisation and 7 days of immobilisation will be used to calculated a fractional synthetic rate (% day).
Change in skeletal muscle gene expression | After 2 days of immobilisation
  Skeletal muscle gene expression will be measured before and after 2 days of single leg immobilisation.
Change in skeletal muscle gene expression | After 7 days of immobilisation
  Skeletal muscle gene expression will be measured before and after 7 days of single leg immobilisation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No